CLINICAL TRIAL: NCT02517983
Title: Phenotyping the Chronic Respiratory Diseases (CRD) in Ho Chi Minh City, Vietnam
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Michel, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-CRD
Record Dates: First submitted 2015-07-28; First posted 2015-08-07 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Respiratory Diseases
Keywords: chronic respiratory diseases phenotyping

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic respiratory disease
  Interventions: Other: epidemiology

INTERVENTIONS:
Other: epidemiology — Relative prevalence of different chronic respiratory disease phenotypes

SUMMARY:
World Health Organization (WHO) considers chronic respiratory disease (CRD) as one of its four priorities. These diseases include asthma and rhinitis, chronic obstructive pulmonary diseases (COPD), occupational lung diseases, sleep apnoea syndromes, pulmonary hypertension, bronchiectasis and interstitial lung diseases. They constitute a serious public health problem in all countries throughout the world, in particular in low and middle income countries and in deprived populations. Hundreds of millions of people of all ages, in all countries of the world, are affected by chronic respiratory diseases. More than 50% of them live in low and middle income countries. Over 90% of deaths and the complete inability, due to CRDs occur in countries with low or middle incomes.

The main causes of CRD are: tobacco smoke, occupational factors, indoor air pollution and outdoor air pollution, allergens, sequelae of respiratory infections such as tuberculosis.

More than 30% of the population of Ho Chi Minh City (HCMC) could develop a CRD. In fact, 15% of children and 7% of adults could become asthma and 6% of the population could become COPD due to smoking. Children exposed to fumes from biomass burning, early in their life, seem to have a higher risk to develop COPD. The high level of air pollution in HCMC could aggravate asthma / COPD. Populations combining the rural risk (exposure to smoke from biomass) and the urban risk (smoking, pollution) may develop COPD much earlier (before age 40). Among the 9 million people in HCMC, 50% of the population is rural origin. Within this population, parasites could play a protective role against the risk of allergic asthma and consequently, the better control of helminthiasis among urban population, may result in allergic diseases such as asthma and anaphylaxis. Finally, the sequelae of tuberculosis (incidence is 200/100000) could participate to the morbidity of COPD / CRD.

Study granted by the ARES-CUD ("Comission universitaire au développement")

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old
* Gender: Female and Male
* Signed informed consent
* Out-patients at the Pham Ngoc Thach Hospital
* One or several symptoms suggesting chronic respiratory disease (cough, chest tightness, wheezing, dyspnoea, sputum), lasting 3 months or more.
* Lung function defect (FEV1/FVC < 0,7 or FEV1 < 80% PV with FEV1/FVC > 0,7 or FEV1> 80% PV and FEV1/FVC > 0,7 with a decrease of DLCO (< 80% PV).

FEV1: Forced Expiratory Volume in 1 Second FVC : Forced Vital Capacity PV: predicted value DLCO: Diffusing Capacity of the Lung for Carbon Monoxide

* Patients are able to stop anti-histamine 5 days before evaluation.
* Patients are able to stop bronchodilator treatment before performing lung function test according to standard practice (immediate release theophylline: 24 hours, long acting β2-agonist: 12 hours, short acting β2-agonist: 6 hours and short acting anticholinergic: 8 hours).

Exclusion Criteria:

* The patients do not agree to participate in the study.
* Presence of one or more chronic diseases: HIV, active tuberculosis, hypertension, heart failure, diabetes, low BMI (<18.5) or mental health disorders.
* Treatment with B-blockers, drugs of vascular/heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The out-patient population with chronic respiratory disease who are admitted in Pham Ngoc Thach Hospital
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Relative prevalence of the different chronic respiratory diseases phenotype | 4 months after start of study
  This will be measured by the percentage of each chronic respiratory diseases phenotype, according to the lung function test.

SECONDARY OUTCOMES:
role of environmental risk factors in developing chronic respiratory diseases | 4 months after start of study
  This will be measured by means of a questionnaire.
role of occupational risk factors in developing chronic respiratory diseases | 4 months after start of study
  This will be measured by means of a questionnaire.
role of clinical risk factors in developing chronic respiratory diseases | 4 months after start of study
  This will be measured by means of a questionnaire and lung function test
Allergen skin reactivity test to assess the role of atopic in developing chronic respiratory diseases | 4 months after start of study
Induced sputum analysis to assess the relationship between phenotype and endotype among a sub-group of chronic respiratory diseases | 4 months after start of study
Biomarkers assessment for risk factors of chronic respiratory diseases | 4 months after start of study
  Total IgE number and specific IgE number if needed depending on each phenotype of chronic respiratory disease

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Michel, MD, Principal Investigator — CHU Brugmann; Ha Chu Thi, MD, Principal Investigator — Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam
Locations (1):
- Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] COPD-more than just tobacco smoke. Lancet. 2009 Aug 29;374(9691):663. doi: 10.1016/S0140-6736(09)61535-X. No abstract available. PMID 19716941
- [Background] Bousquet J, Kiley J, Bateman ED, Viegi G, Cruz AA, Khaltaev N, Ait Khaled N, Baena-Cagnani CE, Barreto ML, Billo N, Canonica GW, Carlsen KH, Chavannes N, Chuchalin A, Drazen J, Fabbri LM, Gerbase MW, Humbert M, Joos G, Masjedi MR, Makino S, Rabe K, To T, Zhi L. Prioritised research agenda for prevention and control of chronic respiratory diseases. Eur Respir J. 2010 Nov;36(5):995-1001. doi: 10.1183/09031936.00012610. Epub 2010 Mar 11. PMID 20223919
- [Background] Flohr C, Tuyen LN, Quinnell RJ, Lewis S, Minh TT, Campbell J, Simmons C, Telford G, Brown A, Hien TT, Farrar J, Williams H, Pritchard DI, Britton J. Reduced helminth burden increases allergen skin sensitization but not clinical allergy: a randomized, double-blind, placebo-controlled trial in Vietnam. Clin Exp Allergy. 2010 Jan;40(1):131-42. doi: 10.1111/j.1365-2222.2009.03346.x. Epub 2009 Sep 15. PMID 19758373
- [Background] Regional COPD Working Group. COPD prevalence in 12 Asia-Pacific countries and regions: projections based on the COPD prevalence estimation model. Respirology. 2003 Jun;8(2):192-8. doi: 10.1046/j.1440-1843.2003.00460.x. PMID 12753535